CLINICAL TRIAL: NCT06758830
Title: Total Neoadjuvant Therapy for Rectal Cancer - a New Standard of Care?
Brief Title: Total Neoadjuvant Therapy and Organ Preservation Versus Surgery for Rectal Cancer.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other)
Collaborators: Vilnius University (Other); Tomas Poskus, Faculty of Medicine, Vilnius University (Unknown); Vilnius University Hospital Santaros Klinikos (Other); Research Council of Lithuania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STart
Record Dates: First submitted 2024-12-19; First posted 2025-01-06 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Rectal Cancer; Total Neoadjuvant Treatment; Neoadjuvant Therapy; Radiotherapy; Chemotherapy; Organ Preservation; Radiotherapy Side Effect; Chemotherapy Side Effects; Chemoradiotherapy; Low Anterior Resection Syndrome; Quality of Life
Keywords: Rectal cancer; Total Neoadjuvant Treatment; Neoadjuvant therapy; Radiotherapy; Chemotherapy; Chemoradiotherapy; Organ Preservation; Radiotherapy Side Effect; Chemotherapy side effects; Quality of Lifte; Fatigue; Postoperative complications; Low Anterior Resection Syndrome
MeSH Terms: conditions — Rectal Neoplasms; Radiation Injuries; Low Anterior Resection Syndrome; Fatigue; Postoperative Complications | interventions — Radiotherapy; Chemoradiotherapy; Consolidation Chemotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: **Part One:** A prospective randomized study. Participants will be randomly divided into two groups: an experimental group and a control group.
  **Part Two:** A prospective cohort study. In the second part of the study, there is no planned allocation of groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part one. The first group: an experimental group - TNT, organ preservation. (Experimental): Participants in the experimental group will be treated with TNT - CRT plus consolidating Ch. Consolidation Ch lasts 12 weeks. The response to TNT will be assessed 4 to 5 weeks after the last cycle of Ch. Response assessment will be performed through digital examination, pelvic MRI, rectoscopy, and biopsy. Participants will be actively followed up and not treated after a complete or near-complete response. In case of non-response, participants will undergo surgery. If the participant is diagnosed with a near-complete clinical response and wishes to avoid surgery, the response is reassessed after 8 weeks. If there is no response, i.e., near-complete clinical response persists, the participant is offered surgery.
  Participants in the experimental group do not receive adjuvant treatment after TNT and surgery.
  Interventions: Radiation: Radiation Therapy; Drug: Chemoradiotherapy; Drug: Consolidation Chemotherapy; Procedure: Surgery
- Part one. Second Group: a control Group - surgery (Active Comparator): In the control group, treatment will start with surgery. Following surgical treatment, adjuvant therapy may be provided for control group participants according to standard clinical practice if indicated.
  Interventions: Procedure: Surgery; Other: Adjuvant treatment
- Part two of the study (Other): In the second part of the study, investigators will prospectively collect and analyze the personal medical records of participants who have already received treatment with CRT or TNT. No new diagnostic or therapeutic approaches will be implemented; routine clinical practices for long-term follow-up will continue. For participants who have not received specific treatment and do not meet the inclusion criteria for the first part of the study, as well as those who declined to participate in that part, investigators will follow the routine clinical practices for investigation, treatment, and follow-up as long as they meet the inclusion criteria for the second part of the study.
  Interventions: Other: Part two

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy (RT) is administered at a dose of 2 Gy per day for a total dose of 50 Gy delivered to the pelvis. This is done throughout 5 to 6 weeks.
  Arms: Part one. The first group: an experimental group - TNT, organ preservation.
Drug: Chemoradiotherapy — Capecitabine: 825 mg/m² twice daily, prescribed 1-5 days per week, for 5 weeks during RT.
  Or Bolus 5-FU regimen: 5-fluorouracil (5-FU) 400 mg/m2/day intravenously, administered on days 1-4 and 33-35. Calcium folinate (folinic acid) 20 mg/m2/day intravenously on days 1-4 and 33-35.
  Arms: Part one. The first group: an experimental group - TNT, organ preservation.
Drug: Consolidation Chemotherapy — XELOX: Oxaliplatin 130 mg/m² (day 1) + capecitabine 1000 mg/m² (days 1-14), every 3 weeks for 4 cycles.
  Or FOLFOX: Oxaliplatin - 85 mg/m2 intravenously (2-hour infusion), drip for 1 day. Calcium folinate (folinic acid) - 400 mg/m2/d. intravenously (2-hour infusion), started on day 1. F(5-fluorouracil) - 400 mg/m2/d. intravenously (bolus), started on day 1. Repeat every 2 weeks for 6 times.
  Arms: Part one. The first group: an experimental group - TNT, organ preservation.
Procedure: Surgery — Transabdominal Resection: Abdominoperineal resection, low anterior resection, or coloanal anastomosis using total mesorectal excision.
  Arms: Part one. Second Group: a control Group - surgery; Part one. The first group: an experimental group - TNT, organ preservation.
Other: Part two — Standard treatment protocols and follow-up procedures are implemented in clinical practice.
  Arms: Part two of the study
Other: Adjuvant treatment — If indicated, adjuvant therapy will be administered as usual in clinical practice.
  Arms: Part one. Second Group: a control Group - surgery

SUMMARY:
This study hypothesizes that approximately 50% of rectal cancer patients can preserve their rectum using a watch-and-wait strategy if they achieve a complete or near-complete clinical response to total neoadjuvant therapy (TNT). The objective is to determine whether the complications, quality of life, and survival rates of rectal cancer patients who have achieved a complete or near-complete clinical response to TNT, followed by a watch-and-wait approach, are comparable to those of patients who undergo surgery first. Additionally, the study aims to identify potential prognostic and predictive markers for rectal cancer and examine survival rates and factors influencing responses to chemoradiotherapy (CRT) or TNT.

The study is divided into two parts:

**Part One:** Participants with cT1N1, T2-T3 N0-1 rectal cancer, MRF-, and EMVI-, with surgery as one of the possible first-line treatment options, will be randomized into two groups. The experimental group will consist of participants receiving TNT, including CRT and consolidation chemotherapy (Ch). If these participants achieve a complete or near-complete clinical response, they will be observed using a watch-and-wait strategy, which is a non-operative approach. The control group will consist of participants who undergo surgical treatment initially.

**Part Two:** All participants with rectal cancer who have received CRT or TNT will be included. Additionally, participants diagnosed with rectal cancer who are scheduled for CRT or TNT but declined to participate in Part One or do not meet the inclusion criteria will also be included.

ELIGIBILITY:
Part One

Inclusion Criteria:

* Over 18 years of age.
* Participants who agreed to participate in the study signed an informed consent form.
* The Eastern Cooperative Oncology Group (ECOG) score ranges from 0 to 2.
* Pathologically confirmed rectal adenocarcinoma.
* Tumor up to 10 cm from the anus.
* Magnetic resonance imaging (MRI) of the pelvis and computed tomography (CT) of the thorax and abdomen were performed to confirm the diagnosis.
* cT1N1, T2-T3 N0 - 1, M0, MRF -, EMVI -.
* Normal bone marrow function: blood leucocytes > 3.5 × 10⁹/l, neutrophils > 1.5 × 10⁹/l, platelets > 100 × 10⁹/l.
* Normal renal function: creatinine within 1,5 × normal.
* Normal liver function: blood bilirubin levels within 1,5 times normal, AST, ALT levels within 2,5 times the upper limit.

Exclusion Criteria:

* Prior ST or Ch.
* Participants who are not eligible for pelvic MRI.
* Participants who have had a malignancy in the last 5 years, except for treatment for basal cell or squamous cell skin cancer or in situ cervical cancer.
* ECOG status ≥ 3.
* Distant metastases detected.
* Participants with uncontrolled therapeutic or psychiatric conditions.
* Infectious diseases requiring antibiotic treatment.

Part Two

Inclusion Criteria:

* Over 18 years of age.
* Participants who agreed to participate in the study signed an informed consent form.
* ECOG score between 0 and 2.
* Pathological confirmed rectal adenocarcinoma.
* Stage I to III rectal cancer confirmed.
* The tumor is localized up to 12 cm from the anus.
* Participants who refused to participate in the first part of the study or did not meet the inclusion criteria for the first part.
* Participants have received preoperative CRT or TNT or are in the planning stages of neoadjuvant treatment.

Exclusion Criteria:

* New cancer two years after CRT.
* Stage IV cancer before treatment.
* Participants refusing to participate in the study or unable to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-07 (Estimated); Primary Completion 2029-12-27 (Estimated); Study Completion 2029-12-27 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | From the start of treatment until 3 months after surgery.
  Assessed based on the Clavien Dindo classification.
TNT toxicity | From the start of treatment until 3 months after TNT.
  Local and systemic toxicity and (or) side effects will be recorded according to the general terminology criteria for adverse events version 5.0 (CTCAE v5.0).
Mortality rate | From the start of treatment until 3 months after treatment.
  Mortality after TNT or surgery.
Quality of life | From the start of treatment until 3 years after treatment.
  Quality of life Will be assessed using scoring manual of European Organisation For Research And Treatment Of Cancer of CR29 (Colorectal).
Low anterior resection syndrome rate. | From the start of treatment until 3 years after treatment.
  Assessed based on the LARS questionnaire
Fatigue | From the start of treatment until 3 years after treatment
  Fatigue will be assessed using scoring manual of the functional assessment of chronic illness therapy - fatigue (FACIT-F) questionnaire.
Complete clinical response rate | 12 - 14 weeks after TNT
  Criteria for Complete Clinical Response
  DRE:
  * Smooth, flat scar
  * No nodularity
  Endoscopy:
  * Pale smooth scar with or without telangiectasia
  * No ulceration, nodularity, or mucosal irregularities
  * No stricture
  MRT:
  * Fibrotic, linear scar with low signal intensity on T2-weighted images
  * No diffusion restriction
  * No suspicious lymph nodes All of the criteria must be satisfied to define a complete clinical response.
Near-complete clinical response rate | 12 - 14 weeks after TNT
  Near Complete Response
  DRE:
  - Smooth induration or superficial minor mucosal irregularity
  Endoscopic:
  * Appearance with irregular small mucosal nodules, superficial ulceration, or mild persistent erythema MRI
  * Downstaging with or without residual fibrosis, small area of residual signal, and complete or partial regression of lymph nodes
  * Diffusion-weighted MRI with a small area of residual high signal intensity

SECONDARY OUTCOMES:
Rectal preservation rate | 3 years after TNT
  Percentage of participants achieving complete or near-complete clinical response and rectal preservation using a "watch and wait" approach.
Local regrowth rate | 3 years after TNT
  Percentage of participants with tumor regrowth after watch-and-wait when a complete or near-complete clinical response was achieved after TNT
Overall survival | 3 - 5 years.
  The time between enrolment and death from any cause.
Disease-free survival | 3 - 5 years.
  The time between enrolment and the first documented disease progression, i.e. local recurrence or metastasis, or death from any cause.
Local recurrence-free survival | 3 - 5 years.
  Local recurrence rates in participants who underwent surgery.
Distant metastasis-free survival | 3 - 5 years.
  Incidence of distant metastases
Stoma free survival | 3 - 5 years.
  Stoma-free survival is defined as the period after treatment during which the patient does not develop a stoma.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Poškus, PhD, Study Chair — Translational Health Research Institute, Faculty of Medicine, Vilnius University Ciurlionio str. 21, LT-03101 Vilnius; Audrius Dulskas, PhD, Principal Investigator — General and Abdominal Surgery and Oncology Department, National Cancer Institute, Vilnius, Lithuania
Locations (1):
- Nacional Cancer Institute, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided